CLINICAL TRIAL: NCT02405078
Title: Pilot Project for Creation of the DLBCL Response Prediction Model: Combining Early Interim Functional Imaging, Detection of a Tumor-Specific Clonotype and Metabolic Profiling of Blood of in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma to Predict Response to Standard Immunochemotherapy
Brief Title: Tumor-Specific Clonotype, Metabolic Profile, and PET/CT in Predicting Chemotherapy Response in Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-0022; NCI-2015-01946 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0022 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Drug Therapy; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (PET/CT, clonotype, metabolic profile) (Experimental): Patients receive standard salvage chemotherapy as determined by the treating physician.
  Patients undergo FDG PET/CT scans at baseline (between days -21 to 0), on day 4 after completion of first high-dose chemotherapy, on day 21 after completion of the first course of chemotherapy, and on day 42 after the end of the second course of chemotherapy. Blood samples are also collected for tumor-specific clonotype and metabolic profile at baseline (days -5 to 0) and on days 4, 8, 21, and 42.
  Interventions: Drug: Chemotherapy; Procedure: Computed Tomography; Drug: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Chemotherapy — Given standard salvage chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Procedure: Computed Tomography — Undergo FDG-PET/CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Drug: Fludeoxyglucose F-18 — Undergo FDG-PET/CT scan
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Positron Emission Tomography — Undergo FDG-PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This pilot clinical trial studies tumor-specific markers (clonotype), blood tests, and positron emission tomography (PET)/computed tomography (CT) in predicting treatment response at different times during chemotherapy in patients with diffuse large B-cell lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Studying samples of blood in the laboratory from patients during chemotherapy may help doctors learn more about the effects of treatment on cells and may help doctors determine whether patients are responding to treatment. PET/CT scan procedures are done at the same time with the same machine and the combined scans give more detailed pictures of areas inside the body than either scan gives by itself and may help doctors find out how well treatment is working.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the ability of blood based detection of a tumor-specific clonotype and metabolic profiling and functional imaging to predict response to standard immunochemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate the optimal time points to create the diffuse large B-cell lymphoma (DLBCL) response prediction model.

TERTIARY OBJECTIVES:

I. To evaluate the prognostic value of clinical factors, cell of origin subtype, and circulating immune cell subsets for response to therapy.

II. To evaluate for novel genomic aberrations or signatures which correlate with therapeutic failure.

III. To evaluate the ability of additional positron emission tomography (PET)/computed tomography (CT) imaging interpretation techniques to correlate with clinical outcomes.

IV. To evaluate the correlation of blood-based detection of clonotype with fludeoxyglucose F-18 (FDG) PET/CT disease assessment.

V. To evaluate the utility of alternative methods of minimal residual disease detection.

VI. To evaluate measurement of circulating metabolic profiling with imaging results and clinical outcomes.

OUTLINE:

Patients receive standard salvage chemotherapy as determined by the treating physician.

Patients undergo FDG PET/CT scans at baseline (between days -21 to 0), on day 4 after completion of first high-dose chemotherapy, on day 21 after completion of the first course of chemotherapy, and on day 42 after the end of the second course of chemotherapy. Blood samples are also collected for tumor-specific clonotype and metabolic profile at baseline (days -5 to 0) and on days 4, 8, 21, and 42.

ELIGIBILITY:
Inclusion Criteria:

* Subject/legal representative willing and able to provide written informed consent
* Histologically confirmed aggressive B-cell DLBCL, including follicular lymphoma (FL) transforming to DLBCL and high grade B-cell lymphoma
* Willing to provide existing relapse-confirmatory DLBCL tumor sample
* Relapsed from or refractory to at least one treatment containing a CD20 monoclonal antibody combined with anthracycline-based chemotherapy
* CT scans showing involvement of 1 or more clearly demarcated lesions with a long axis > 1.5 cm and short axis >= 1.0 cm
* Baseline FDG-PET/CT scans must demonstrate at least one hypermetabolic lesion as defined by the Deauville criteria localizing to CT-defined anatomical tumor sites
* Suitable candidate for therapy with standard salvage chemotherapy and autologous stem cell transplant (ASCT) as determined by the treating physician
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy of >= 12 weeks as estimated by the treating physician
* Negative serum beta-human chorionic gonadotropin (beta-hCG) test (women of childbearing potential only)
* Hemoglobin >= 8.5 g/dL
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 75,000/mm^3
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 5 x institutional upper limit of normal (ULN) for cases involving liver metastasis and =< 3 x institutional ULN for all other cases
* Bilirubin =< 2 x ULN (unless related to lymphoma) or =< 5 x ULN for subjects with documented or suspected Gilbert's disease
* Serum creatinine =< 1.5 x ULN or calculated creatinine clearance (CrCl) >= 50 mL/min as determined by the Cockcroft-Gault equation

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, would interfere with the interpretation of study results or subject safety including non-malignant FDG avid diseases such as sarcoidosis or other granulomatous disease
* Uncontrolled diabetes mellitus
* Concurrent enrollment in another clinical study where they are receiving non-standard salvage chemotherapy, (i.e., concurrent enrollment is allowable if the patient is receiving standard salvage chemotherapy and research imaging is allowed)
* Any chemotherapy, radiotherapy, immunotherapy, biologic, or investigational therapy for treatment of lymphoma within 14 days prior to treatment
* Symptomatic congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Response to therapy | Up to 42 days
  Defined as demonstrating the chemotherapy-sensitiveness for curative autologous stem cell transplant (ASCT) based on fludeoxyglucose F 18 FDG positron emission tomography (PET)/computed tomography (CT) results. Non-responders will be classified as having equivocal active disease with a positive biopsy for confirmation and unequivocal active disease in a previously biopsy-confirmed site of disease. Descriptive statistics will be used to summarize the demographic and clinical characteristics of patients. The concordance rate between the interim PET/CT scans and the final FDG PET/CT scan, and its 95% confidence interval, will be reported. The change in drug of choice (DoC) and metabolic profile tests will be explored using mixed effect linear regression models.

SECONDARY OUTCOMES:
Response rate (RR) | Up to 18 months
  RR will be analyzed using multivariate logistic regression.
Progression-free survival | Up to 18 months
  The association between FDG PET/CT scans, DoC and metabolic profile tests, and the progression-free from primary treatment failure will be examined using a stratified Cox regression model.
Overall survival (OS) | Up to 18 months
  The association between FDG PET/CT scans, DoC and metabolic profile tests, and the OS from primary treatment failure will be examined using a stratified Cox regression model.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Westin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Cherng HJ, Chuang HH, Steiner R, Fayad L, Strati P, Nair R, Hagemeister F, Nastoupil LJ, Lee HJ, Neelapu SS, Flowers CR, Samaniego F, Rodriguez M, Macapinlac HA, Feng L, Westin J. A prospective study on early PET/CT scans during the first cycle of salvage chemotherapy for relapsed or refractory diffuse large B-cell lymphoma. Leuk Lymphoma. 2022 Jan;63(1):74-83. doi: 10.1080/10428194.2021.1971223. Epub 2021 Aug 26. PMID 34435552
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org